CLINICAL TRIAL: NCT01910597
Title: Phase I, Dose-Escalation Study of Soluble Beta-Glucan (SBG) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Arunee Dechaphunkul, Dr, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 552941411
Record Dates: First submitted 2013-07-23; First posted 2013-07-29 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBG (Experimental)
  Interventions: Drug: SBG

INTERVENTIONS:
Drug: SBG

SUMMARY:
Soluble Beta-Glucan (SBG) is a compound prepared from commercial active dry Baker's yeast which is then proceeded through a multi-step laboratory processes invented by Prof. Rapepun Wititsuwannakul, Faculty of Science, Prince of Songkla University, Thailand. Based upon pre-clinical data, SBG has been shown to inhibit angiogenesis and probably enhance immune function, leading to shrinkage of tumor size in athymic nude mice injected by hepatocellular carcinoma cells (HepG2) and cervical cancer cells. Therefore, the investigators expect to see the safety and anti-cancer property of SBG in patients with advanced cancer whom no available therapy can be offered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically documented, advanced-stage, primary or metastatic solid tumors that are refractory to standard therapy or for which no available standard therapy exists.
* Evidence of measurable or evaluable disease.
* Age must be at least 18 years.
* ECOG performance status must be 0 or 2.
* Received only best supportive care.
* Patient must meet protocol-specified laboratory values.

Exclusion Criteria:

* Second primary cancer diagnosed within 5 years, except cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma which completed curative treatment.
* Concurrent therapy with any other investigational agent.
* Severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study-drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, make the subject inappropriate for this study.
* Allergy to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) to define the maximum tolerated dose (MTD). The DLT is defined as treatment related grade 3 or grade 4 adverse events or abnormal lab test that occurred in the first 28 days after start of study drug. | continuous monitoring for the first 28 days after start of the study medication

SECONDARY OUTCOMES:
Antitumor activity by comparing baseline and post-treatment changes. Tumor assessment will be performed using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | baseline, month 2, month 4, month 6 and month 8
  baseline and then once every 2 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Arunee Dechaphunkul, MD, Principal Investigator — Prince of Songkla University, Thailand
Locations (1):
- Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand